CLINICAL TRIAL: NCT01103882
Title: Short-Term Clinical Outcome Including Dislocation Rate and Ceramic Fracture of Total Hip Arthroplasty Using Larger Diameter of 4th Generation Ceramic Bearing
Brief Title: Short-Term Clinical Outcome of Total Hip Arthroplasty Using Larger Diameter of 4th Generation Ceramic Bearing
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: INT.CR.LKR1.10
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Arthropathy of Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of this clinical study include:

* Assess the rate of dislocation and fracture of THA using the new (the 4th generation) ceramic implants.
* Evaluate the survival rate of THA using the new alumina-zirconia (the 4th generation) composite ceramic bearing.
* Investigate the performance of the 4th generation ceramic implants mostly in patients younger than 50 years.
* Compare the preoperative and postoperative scores of Harris Hip Score, UCLA Activity Score and WOMAC.

DETAILED DESCRIPTION:
This study will evaluate incidence of dislocation and short-term clinical outcome on patients who undergo large diameter 4th generation ceramic bearing total hip Arthroplasty ("THA") in comparison to historical data on 3rd generation CoC THA (28mm) patients. Specifically the study intends to address the following research topics:

1. The incidence of dislocation after THA with use of the 4th generation Ceramic Bearing in comparison to 3rd generation Ceramic Bearing.
2. The incidence of ceramic fracture after THA with use of the 4th generation Ceramic Bearing in comparison to 3rd generation Ceramic Bearing
3. The survival rate, wear rate, and incidence of osteolysis of THA with use of the 4th generation Ceramic Bearing
4. Range of motion improvement from preoperative to postoperative to support Korean sitting style after THA with use of the 4th generation Ceramic Bearing.
5. Clinical outcomes, activity level and QoL of patients with use of the 4th generation Ceramic Bearing.
6. The performance of THA with use of the new ceramic bearing mostly in patients younger than 50 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for primary Total Hip Replacement
* Patients with degenerative joint disease (inflammatory or non-inflammatory) or any of the composite diagnoses of:

  1. Osteoarthritis
  2. Avascular necrosis
  3. Legg Perthes
  4. Rheumatoid Arthritis
  5. Diastrophic variant
  6. Fracture of the pelvis
  7. Fused hip
  8. Slipped capital epiphysis
  9. Subcapital fractures
  10. Traumatic arthritis
* Patients aged over 20
* Patients must be able to understand instructions and be willing to return for follow-up

Exclusion Criteria:

* Absolute contraindications include: infection, sepsis, and osteomyelitis
* Relative contraindications include:

  1. uncooperative patient or patient with neurologic disorders who are incapable of following directions,
  2. osteoporosis,
  3. metabolic disorders which may impair bone formation,
  4. osteomalacia,
  5. distant foci of infections which may spread to the implant site,
  6. rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram, and
  7. vascular insufficiency, muscular atrophy, or neuromuscular disease.
  8. pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for total hip arthroplasty
Sampling Method: Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Dislocation | 12 month postop
  Number of dislocations

SECONDARY OUTCOMES:
Clinical Outcomes | 12 months, 18 months and 30 months
  Harris Hip Score, UCLA and WOMAC

CONTACTS AND LOCATIONS:
Overall Officials: Woon-Hwa Jung, M.D., Principal Investigator — Murup Hospital, Masan, Korea; Yong-Chan Ha, M.D., Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Yong-Kyun Lee, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Tae-Young Kim, M.D., Principal Investigator — Hallym University Hospital
Locations (4):
- South Korea (4):
  - Hallym University Hospital, Anyang
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Murup Hospital, Masan
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No